CLINICAL TRIAL: NCT04997148
Title: Cladribine Tablets in Highly-active Relapsing Multiple Sclerosis - Real-World Effectiveness in UK Clinical Practice (CAMELOT-MS)
Brief Title: Effectiveness of Cladribine Tablets in Participants With Highly-active Relapsing Multiple Sclerosis (CAMELOT-MS)
Status: Completed | Type: Observational
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Limited, UK (Industry)
Responsible Party: Sponsor
Other Study IDs: MS700568_0150
Record Dates: First submitted 2021-08-03; First posted 2021-08-09 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Mavenclad ®; Cladribine
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cladribine: No intervention was administered as a part of this study. Participants with Highly-active Disease Relapsing-remitting Multiple Sclerosis (HDA-RRMS), who completed at least Year 1 of treatment with cladribine tablets in routine clinical practice were enrolled into this study and assessed up to maximum 5 years after cladribine tablets initiation.

SUMMARY:
The main purpose of this study was to investigate the effectiveness of cladribine tablets in a UK real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of HDA-RRMS as defined by clinical or radiological features
* Treatment initiation with cladribine tablet monotherapy on or after 22 August 2017 and at least 3 years before enrolment
* Completion of Year 1 treatment of cladribine tablets (Week 1 and Week 2 treatment, per recommended dose in Year 1: 1.75 milligrams per kilogram [mg/kg] body weight, cumulatively)

Exclusion Criteria:

* Received cladribine tablet treatment within an interventional clinical trial during the study period
* Received treatment with any investigational therapy for RRMS in the 6 months prior to cladribine tablet treatment initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with HDA-RRMS who initiated treatment with cladribine tablets.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (8):
- United Kingdom (8):
  - University Hospitals Coventry and Warwickshire- Neurology, Coventry
  - NHS Lanarkshire Health Board- Department of Neurology, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - University Hospitals of Leicester NHS Trust, Leicester
  - Barking Havering and Redbridge University Hospitals NHS Trust, London
  - University College London UCL, London
  - Nottingham City Hospital (2655), Nottingham
  - Salford Royal, Salford

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS700568_0150
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cladribine: Participants diagnosed with Highly-active Disease Relapsing-remitting Multiple Sclerosis (HDA-RRMS), who completed at least Year 1 of treatment with cladribine tablets in routine clinical practice were enrolled into this study and assessed up to maximum 5 years after cladribine tablets initiation.
Period: Overall Study
Arm/Group | Cladribine
Started | 116
Completed | 116
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cladribine
Number analyzed (Participants) | 116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 116

OUTCOME MEASURES:

1. Secondary Outcome: Relapse-Free Rate in Each Year After Initiation of Cladribine Tablet Treatment
Description: Relapse-free is defined as the time from the on-treatment period start date until first relapse or death as assessed by the investigator. Relapse-free rate, i.e., the survival rate using Kaplan Meier method, was summarized every year.
Time Frame: Year 1, 2, 3, 4 and 5 after treatment initiation with Cladribine tablets until relapse or death
Population: Full Analysis Set included all participants who were treated with at least one course of treatment with cladribine tablets. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at specified time points for this outcome measure.
Measure: Number (95% Confidence Interval); unit: estimated probability
Arm/Group | Cladribine
Number analyzed (Participants) | 116
estimated probability
  Year 1 | 0.92 [0.80 to 0.97]
  Year 2 | 0.85 [0.72 to 0.93]
  Year 3 | 0.81 [0.67 to 0.90]
  Year 4 | 0.78 [0.63 to 0.87]
  Year 5 | 0.75 [0.58 to 0.86]

2. Primary Outcome: Annualized Relapse Rate in the Year Prior to Treatment Initiation With Cladribine Tablets
Description: The annualized relapse rate for a participant is defined here as the number of clinician's confirmed relapses that occurred in the year prior to the date of Cladribine tablet initiation.
Time Frame: 1 Year prior to date of Cladribine tablet initiation
Population: Full Analysis Set included all participants who were treated with at least one course of treatment with cladribine tablets.
Measure: Mean (95% Confidence Interval); unit: Relapse per year
Arm/Group | Cladribine
Number analyzed (Participants) | 116
Relapse per year | 0.595 [0.470 to 0.753]

3. Primary Outcome: Annualized Relapse Rate in the Year One After Treatment Initiation With Cladribine Tablets
Description: The annualized relapse rate for a participant is defined here as the number of clinician's confirmed relapses that occurred in Year 1 after treatment initiation with Cladribine tablets.
Time Frame: Year 1 after treatment initiation with Cladribine tablets
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Relapse per year
Arm/Group | Cladribine
Number analyzed (Participants) | 116
Relapse per year | 0.101 [0.052 to 0.194]

4. Primary Outcome: Annualized Relapse Rate in the Year 2 After Treatment Initiation With Cladribine Tablets
Description: The annualized relapse rate for a participant is defined here as the number of clinician's confirmed relapses that occurred in Years 2 after treatment initiation with Cladribine tablets.
Time Frame: Year 2 after treatment initiation with Cladribine tablets
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Relapse per year
Arm/Group | Cladribine
Number analyzed (Participants) | 116
Relapse per year | 0.052 [0.023 to 0.115]

5. Primary Outcome: Annualized Relapse Rate in the Year 3 After Treatment Initiation With Cladribine Tablets
Description: The annualized relapse rate for a participant is defined here as the number of clinician's confirmed relapses that occurred in Year 3 after treatment initiation with Cladribine tablets.
Time Frame: Year 3 after treatment initiation with Cladribine tablets
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Relapse per year
Arm/Group | Cladribine
Number analyzed (Participants) | 116
Relapse per year | 0.086 [0.046 to 0.160]

6. Primary Outcome: Annualized Relapse Rate in the Year 4 After Treatment Initiation With Cladribine Tablets
Description: The annualized relapse rate for a participant is defined here as the number of clinician's confirmed relapses that occurred in Years 4 after treatment initiation with Cladribine tablets.
Time Frame: Year 4 after treatment initiation with Cladribine tablets
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Relapse per year
Arm/Group | Cladribine
Number analyzed (Participants) | 116
Relapse per year | 0.060 [0.046 to 0.160]

7. Primary Outcome: Annualized Relapse Rate in the Year 5 After Treatment Initiation With Cladribine Tablets
Description: The annualized relapse rate for a participant is defined here as the number of clinician's confirmed relapses that occurred in Year 5 after treatment initiation with Cladribine tablets.
Time Frame: Year 5 after treatment initiation with Cladribine tablets
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Relapse per year
Arm/Group | Cladribine
Number analyzed (Participants) | 116
Relapse per year | 0.063 [0.024 to 0.169]

8. Secondary Outcome: Time From Cladribine Tablet Initiation to First Relapse
Description: A qualifying relapse is defined as new, worsening or recurrent neurological symptoms attributed to Multiple Sclerosis (MS) that last for at least 24 hours without fever or infection, or adverse reaction to prescribed medication, preceded by a stable or improving neurological status of at least 30 days. Percentage of participants with qualified relapse-free status at week 24 were reported.
Time Frame: up to maximum 5 years after treatment initiation with Cladribine tablets
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Cladribine
Number analyzed (Participants) | 116
years | NA [NA to NA] — Median time to relapse and CI was not reached due to insufficient number of participants with events.

9. Secondary Outcome: Number of Participants Who Discontinued Cladribine Tablets
Description: The number of participants who discontinued treatment with cladribine are reported here.
Time Frame: From Cladribine treatment initiation up to end of Cladribine treatment (assessed up end of Treatment Year 2)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine
Number analyzed (Participants) | 116
Participants | 4

10. Secondary Outcome: Number of Participants Who Received Subsequent Disease-modifying Therapies (DMTs) After Cladribine Tablets Discontinuation/Treatment Completion
Description: The number of participants who received Subsequent Disease-modifying Therapies (DMTs) after Cladribine Tablets Discontinuation/Treatment Completion were reported here.
Time Frame: From Cladribine treatment initiation up to end of Cladribine treatment (assessed up end of Treatment Year 2)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine
Number analyzed (Participants) | 116
Participants | 19

11. Secondary Outcome: Number of Participants With Disability Progression Assessed by Expanded Disease Severity Scale (EDSS) at Treatment Initiation and Start of Treatment Year 2
Description: he EDSS is an ordinal clinical rating scale in half-point increments. It assesses the following eight functional systems, areas of the central nervous system that control bodily functions: Pyramidal (ability to walk), Cerebellar (coordination), Brain stem (speech and swallowing), Sensory (touch and pain), Bowel and bladder functions, Visual, Mental, Other (includes any other neurological findings due to Multiple Sclerosis [MS]). EDSS overall score ranging from 0 (normal) to 10 (death due to MS).
Time Frame: At Treatment Initiation and Start of Treatment Year 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine
Number analyzed (Participants) | 116
Participants | 0

12. Secondary Outcome: Number of Participants With Disability Progression Confirmed Over 6 Months, Assessed by Expanded Disease Severity Scale (EDSS) at 2 Years After Cladribine Tablet Treatment Initiation
Description: as for outcome 11
Time Frame: At 2 years after treatment initiation with Cladribine tablets
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine
Number analyzed (Participants) | 116
Participants | 0

13. Secondary Outcome: Number of Participants With Grade 3 Lymphopenia, Grade 4 Lymphopenia, Herpes Infections, Serious Infections, Opportunistic Infections and Malignancies
Description: Number of Participants with Grade 3 Lymphopenia, Grade 4 Lymphopenia, Herpes Infections, Serious Infections, Opportunistic Infections and Malignancies were reported.
Time Frame: At 2 years after treatment initiation with Cladribine tablets
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine
Number analyzed (Participants) | 116
Participants
  Grade 3 Lymphopenia | 47
  Grade 4 Lymphopenia | 0
  Herpes infections | 6
  Serious/opportunistic infections | 8
  Malignancies | 1

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Cladribine
All-Cause Mortality (participants affected / at risk) | 0/116
Serious Adverse Events (participants affected / at risk) | 1/116
Other Adverse Events (participants affected / at risk) | 51/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cladribine (N=116)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cladribine (N=116)
Lymphopenia (Blood and lymphatic system disorders) | 47 (47)
Herpes simplex (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)

LIMITATIONS AND CAVEATS:
Potential limitations include the retrospective study design, and that data was limited by control over patient assessment as patient monitoring and diagnostics were per standard of care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT04997148/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT04997148/SAP_001.pdf